CLINICAL TRIAL: NCT05833269
Title: Diseño, Implementación Y Evaluación De Un Programa De Intervención Basado En Prácticas De Mindfulness Para El Abordaje Del "burnout Parental" En Mamás Que Realizan Teletrabajo
Brief Title: Intercare, Mindfulness and Compassion Based Intervention for Parental Burnout
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Diego Portales (Other)
Collaborators: Instituto de Seguridad del Trabajo, Chile (Unknown)
Responsible Party: Principal Investigator, Francisco Javier Villalon Lopez, Principal Invesigator, University Diego Portales
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 38-2022
Record Dates: First submitted 2023-04-06; First posted 2023-04-27 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-09

CONDITIONS: Parental Burnout; Burnout, Caregiver; Burnout
Keywords: Parental Burnout; Burnout; Mindfulness; Compassion; Intercare
MeSH Terms: conditions — Caregiver Burden; Burnout, Psychological | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mindfulness and compassion based intercare program (Experimental): This 8-week intervention aims to reduce parental burnout by adapting the "Mindfulness-based Inter-care Program" and incorporating elements from MBSR, MBCT, and CBCT. The program includes 8 modules with practical and theoretical activities, weekly tasks, journaling, and daily meditation practices such as body exploration, seated and moving meditation, walking and eating meditation, acceptance, compassion, and gratitude.
  The program also promotes values such as time management, attentive parenting, and emotional management while addressing factors of risk for parental burnout such as perfectionism, low emotional intelligence, lack of parenting practices, excessive responsibilities, and lack of support. Participants will receive two weekly reminders via email to perform the practices and review information. Additionally, they will have the option to participate in a virtual group via the WhatsApp platform with other participants.
  Interventions: Behavioral: Mindfulness and Compassion based Intercare program for parental burnout reduction (IBAP-BP); Behavioral: Educational material; Behavioral: Reminder by email; Behavioral: Whatsapp support group; Behavioral: Journaling
- Audio guide relaxation control group (Active Comparator): The active control group in this study will be provided with a 20-minute relaxation audio containing Jacobson's progressive relaxation instructions. This intervention aims to control for attention and time while allowing for comparison to the experimental group. Also, journaling was included.
  Additionally, the program will include information on risk factors for parental burnout, such as parental perfectionism, low emotional intelligence, lack of parenting practices, excessive responsibilities, and lack of support. Two weekly email reminders will be sent to encourage daily practice and review of the information provided. Participants will also have the option to participate in a virtual support group through the WhatsApp platform with other participants. This active control group intervention aims to improve participant well-being by providing relaxation techniques and support for the challenges of parenting.
  Interventions: Behavioral: Educational material; Behavioral: Reminder by email; Behavioral: Whatsapp support group; Behavioral: Journaling; Behavioral: Guided relaxation excercise
- Waiting List Group (No Intervention): The waiting list group will receive the intervention after the primary outcome is measured. No intervention was provided before this point.

INTERVENTIONS:
Behavioral: Mindfulness and Compassion based Intercare program for parental burnout reduction (IBAP-BP) — The interventions is an adaptation of an 8-week program called Mindfulness and Compassion based Intercare program designed to reduce burnout. The adaptation includes a parental burnout risk and resource balance framework, focusing on factors such as parental perfectionism, low emotional intelligence, lack of parenting practices, excess parental responsibilities, lack of co-parental support, and lack of social support. The program consists of 8 modules with practical and theoretical activities and daily tasks that require 10-30 minutes. The modules cover topics such as mindfulness, coping with stress, empathy, and self-care. Formal meditation practices include body exploration, sitting, movement, walking, eating, acceptance, compassion, and gratitude. The program also includes descriptions and motivation for practices related to identifying values that promote parenting, time management, attentive parenting techniques, and emotional management.
  Other Names: Intercuidado basado en atencion plena
  Arms: Mindfulness and compassion based intercare program
Behavioral: Educational material — On a weekly basis, participants will receive reminder emails highlighting specific risk factors associated with parental burnout. These risk factors include parental perfectionism, low emotional intelligence, lack of parenting practices, excessive responsibilities, and lack of support. Each week, the reminder email will cover a different topic, providing participants with relevant information.
  Arms: Audio guide relaxation control group; Mindfulness and compassion based intercare program
Behavioral: Reminder by email — Every week, participants will receive two reminder emails: one with a list of activities to complete during the week and another containing information about parental burnout. This approach aims to support participants in staying engaged with the program.
  Arms: Audio guide relaxation control group; Mindfulness and compassion based intercare program
Behavioral: Whatsapp support group — The participants will have the option to join a WhatsApp group with 25 other members from the specific group to receive daily greetings, group support, and have general doubts resolved.
  Arms: Audio guide relaxation control group; Mindfulness and compassion based intercare program
Behavioral: Journaling — As part of the mindfulness intervention, participants are required to write in a journal every day with the purpose of cultivating awareness of bodily sensations, emotions, thoughts, and impulses. Each week, the journaling topic focuses on a different area, including pleasant experiences, unpleasant experiences, needs and resources, communication difficulties, and sharing resources. In contrast, the control group's journaling activity involves free writing about everyday issues, thoughts, and ideas.
  Arms: Audio guide relaxation control group; Mindfulness and compassion based intercare program
Behavioral: Guided relaxation excercise — Participants receive a 10 and 20-minute relaxation exercise guide called the Jacobson Progressive Relaxation, which they are expected to practice daily.
  Arms: Audio guide relaxation control group

SUMMARY:
The goal of this clinical trial is to test the effectiveness of an adapted mindfulness and compassion-based intervention (IBAP) in reducing parental burnout in Chilean mothers who telework while living with children under 18 years old. The main questions it aims to answer are:

* Can the intervention reduce symptoms of parental burnout in the short term (3 months) and medium-term (6 and 9 months) compared to the control group?
* Can the intervention improve work engagement in the intervention group compared to the control group?

Participants will be randomly assigned to either the intervention group or the active control group. The intervention group will receive the IBAP program while the active control group will receive a relaxation audio guide. Both group will receive parental burnout educational material, invitation to a Whatsapp group and a weekly email reminders. Parental Burnout (PBA) will be measured at baseline, 3, 6, and 9 months, and work engagement will be measured at the same time points.

Researchers will compare the intervention group to the active control group to see if the IBM program is more effective in reducing parental burnout and improving work engagement,

ELIGIBILITY:
Inclusion Criteria:

* Mother living with at leat one child over the same roof
* Telework at leat one day per week
* Work at leat three days per week

Exclusion Criteria:

* Self reported acute severe depression
* Self reported psychotic disorder
* Self reported substance abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 250 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Parental Burnout Assessment | 9 months
  The Parental Burnout Assessment (PBA) is a questionnaire validated in Chile that consists of 23 items and evaluates the four main symptoms of parental burnout: emotional exhaustion (9 items), contrast with the parent's previous self (6 items; e.g., I tell myself that I am no longer the parent I used to be), loss of pleasure in the parenting role (5 items; e.g., I don't enjoy spending time with my children), and emotional distancing from children (3 items; e.g., I can no longer show my children that I love them). A 7-point frequency scale is used, with higher scores indicating higher levels of parental burnout. The score is calculated by adding up the scores of the items, with a maximum score of 138 points (Roskam et al., 2021).

SECONDARY OUTCOMES:
Parental Burnout Assessment | 3 months
  The Parental Burnout Assessment (PBA) is a questionnaire validated in Chile that consists of 23 items and evaluates the four main symptoms of parental burnout: emotional exhaustion (9 items), contrast with the parent's previous self (6 items; e.g., I tell myself that I am no longer the parent I used to be), loss of pleasure in the parenting role (5 items; e.g., I don't enjoy spending time with my children), and emotional distancing from children (3 items; e.g., I can no longer show my children that I love them). A 7-point frequency scale is used, with higher scores indicating higher levels of parental burnout. The score is calculated by adding up the scores of the items, with a maximum score of 138 points (Roskam et al., 2021).
Parental Burnout Assessment | 12 months
  The Parental Burnout Assessment (PBA) is a questionnaire validated in Chile that consists of 23 items and evaluates the four main symptoms of parental burnout: emotional exhaustion (9 items), contrast with the parent's previous self (6 items; e.g., I tell myself that I am no longer the parent I used to be), loss of pleasure in the parenting role (5 items; e.g., I don't enjoy spending time with my children), and emotional distancing from children (3 items; e.g., I can no longer show my children that I love them). A 7-point frequency scale is used, with higher scores indicating higher levels of parental burnout. The score is calculated by adding up the scores of the items, with a maximum score of 138 points (Roskam et al., 2021).
Parental Burnout Assessment | 18 months
  The Parental Burnout Assessment (PBA) is a questionnaire validated in Chile that consists of 23 items and evaluates the four main symptoms of parental burnout: emotional exhaustion (9 items), contrast with the parent's previous self (6 items; e.g., I tell myself that I am no longer the parent I used to be), loss of pleasure in the parenting role (5 items; e.g., I don't enjoy spending time with my children), and emotional distancing from children (3 items; e.g., I can no longer show my children that I love them). A 7-point frequency scale is used, with higher scores indicating higher levels of parental burnout. The score is calculated by adding up the scores of the items, with a maximum score of 138 points (Roskam et al., 2021).
Parental Burnout Assessment | 24 months
  The Parental Burnout Assessment (PBA) is a questionnaire validated in Chile that consists of 23 items and evaluates the four main symptoms of parental burnout: emotional exhaustion (9 items), contrast with the parent's previous self (6 items; e.g., I tell myself that I am no longer the parent I used to be), loss of pleasure in the parenting role (5 items; e.g., I don't enjoy spending time with my children), and emotional distancing from children (3 items; e.g., I can no longer show my children that I love them). A 7-point frequency scale is used, with higher scores indicating higher levels of parental burnout. The score is calculated by adding up the scores of the items, with a maximum score of 138 points (Roskam et al., 2021).
Five Facets of Mindfulness Questionnaire - 15 items | 3 months
  The 15-item Five Facets of Mindfulness Questionnaire (FFMQ-15) validated in Chile (Villalon et al, in press) was used.
  The items evaluate the level of certainty of a statement on a Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true), worded both positively and negatively. This questionnaire assesses five dimensions or factors of the mindfulness construct (Observing, Describe, Acting with attention/awareness, Non-judgment of inner experience and Non-reactivity to inner experience). A higher score indicates a higher level of mindfulness.
Five Facets of Mindfulness Questionnaire - 15 items | 6 months
  The 15-item Five Facets of Mindfulness Questionnaire (FFMQ-15) validated in Chile (Villalon et al, in press) was used.
  The items evaluate the level of certainty of a statement on a Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true), worded both positively and negatively. This questionnaire assesses five dimensions or factors of the mindfulness construct (Observing, Describe, Acting with attention/awareness, Non-judgment of inner experience and Non-reactivity to inner experience). A higher score indicates a higher level of mindfulness.
Five Facets of Mindfulness Questionnaire - 15 items | 9 months
  The 15-item Five Facets of Mindfulness Questionnaire (FFMQ-15) validated in Chile (Villalon et al, in press) was used.
  The items evaluate the level of certainty of a statement on a Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true), worded both positively and negatively. This questionnaire assesses five dimensions or factors of the mindfulness construct (Observing, Describe, Acting with attention/awareness, Non-judgment of inner experience and Non-reactivity to inner experience). A higher score indicates a higher level of mindfulness.
Five Facets of Mindfulness Questionnaire - 15 items | 12 months
  The 15-item Five Facets of Mindfulness Questionnaire (FFMQ-15) validated in Chile (Villalon et al, in press) was used.
  The items evaluate the level of certainty of a statement on a Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true), worded both positively and negatively. This questionnaire assesses five dimensions or factors of the mindfulness construct (Observing, Describe, Acting with attention/awareness, Non-judgment of inner experience and Non-reactivity to inner experience). A higher score indicates a higher level of mindfulness.
Five Facets of Mindfulness Questionnaire - 15 items | 18 months
  The 15-item Five Facets of Mindfulness Questionnaire (FFMQ-15) validated in Chile (Villalon et al, in press) was used.
  The items evaluate the level of certainty of a statement on a Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true), worded both positively and negatively. This questionnaire assesses five dimensions or factors of the mindfulness construct (Observing, Describe, Acting with attention/awareness, Non-judgment of inner experience and Non-reactivity to inner experience). A higher score indicates a higher level of mindfulness.
Five Facets of Mindfulness Questionnaire - 15 items | 24 months
  The 15-item Five Facets of Mindfulness Questionnaire (FFMQ-15) validated in Chile (Villalon et al, in press) was used.
  The items evaluate the level of certainty of a statement on a Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true), worded both positively and negatively. This questionnaire assesses five dimensions or factors of the mindfulness construct (Observing, Describe, Acting with attention/awareness, Non-judgment of inner experience and Non-reactivity to inner experience). A higher score indicates a higher level of mindfulness.
Utrecht Work Engagament Scale - 9 | 3 months
  The UWES-9 Spanish version (Schaufeli & Bakker, 2003) was used to assess work engagement. This scale consists of 3 items per dimension, which are vigor, dedication, and absorption (Table 1). Vigor is evaluated through the following 3 items, which refer to high levels of energy and resilience, the willingness to exert effort, not getting tired easily, and persistence in the face of difficulties. Dedication is evaluated through 3 items that refer to the sense or meaning of work, feeling excited and proud of one's work, and feeling inspired and challenged by work. Absorption is evaluated through 3 items that refer to being happily immersed in one's work and having difficulty leaving it, such that time passes quickly and there is forgetfulness of everything else around. The higher the score, the higher the level of work engagement.
Utrecht Work Engagament Scale - 9 | 6 months
  The UWES-9 Spanish version (Schaufeli & Bakker, 2003) was used to assess work engagement. This scale consists of 3 items per dimension, which are vigor, dedication, and absorption (Table 1). Vigor is evaluated through the following 3 items, which refer to high levels of energy and resilience, the willingness to exert effort, not getting tired easily, and persistence in the face of difficulties. Dedication is evaluated through 3 items that refer to the sense or meaning of work, feeling excited and proud of one's work, and feeling inspired and challenged by work. Absorption is evaluated through 3 items that refer to being happily immersed in one's work and having difficulty leaving it, such that time passes quickly and there is forgetfulness of everything else around. The higher the score, the higher the level of work engagement.
Utrecht Work Engagament Scale - 9 | 9 months
  The UWES-9 Spanish version (Schaufeli & Bakker, 2003) was used to assess work engagement. This scale consists of 3 items per dimension, which are vigor, dedication, and absorption (Table 1). Vigor is evaluated through the following 3 items, which refer to high levels of energy and resilience, the willingness to exert effort, not getting tired easily, and persistence in the face of difficulties. Dedication is evaluated through 3 items that refer to the sense or meaning of work, feeling excited and proud of one's work, and feeling inspired and challenged by work. Absorption is evaluated through 3 items that refer to being happily immersed in one's work and having difficulty leaving it, such that time passes quickly and there is forgetfulness of everything else around. The higher the score, the higher the level of work engagement.
Utrecht Work Engagament Scale - 9 | 12 months
  The UWES-9 Spanish version (Schaufeli & Bakker, 2003) was used to assess work engagement. This scale consists of 3 items per dimension, which are vigor, dedication, and absorption (Table 1). Vigor is evaluated through the following 3 items, which refer to high levels of energy and resilience, the willingness to exert effort, not getting tired easily, and persistence in the face of difficulties. Dedication is evaluated through 3 items that refer to the sense or meaning of work, feeling excited and proud of one's work, and feeling inspired and challenged by work. Absorption is evaluated through 3 items that refer to being happily immersed in one's work and having difficulty leaving it, such that time passes quickly and there is forgetfulness of everything else around. The higher the score, the higher the level of work engagement.
Utrecht Work Engagament Scale - 9 | 18 months
  The UWES-9 Spanish version (Schaufeli & Bakker, 2003) was used to assess work engagement. This scale consists of 3 items per dimension, which are vigor, dedication, and absorption (Table 1). Vigor is evaluated through the following 3 items, which refer to high levels of energy and resilience, the willingness to exert effort, not getting tired easily, and persistence in the face of difficulties. Dedication is evaluated through 3 items that refer to the sense or meaning of work, feeling excited and proud of one's work, and feeling inspired and challenged by work. Absorption is evaluated through 3 items that refer to being happily immersed in one's work and having difficulty leaving it, such that time passes quickly and there is forgetfulness of everything else around. The higher the score, the higher the level of work engagement.
Utrecht Work Engagament Scale - 9 | 24 months
  The UWES-9 Spanish version (Schaufeli & Bakker, 2003) was used to assess work engagement. This scale consists of 3 items per dimension, which are vigor, dedication, and absorption (Table 1). Vigor is evaluated through the following 3 items, which refer to high levels of energy and resilience, the willingness to exert effort, not getting tired easily, and persistence in the face of difficulties. Dedication is evaluated through 3 items that refer to the sense or meaning of work, feeling excited and proud of one's work, and feeling inspired and challenged by work. Absorption is evaluated through 3 items that refer to being happily immersed in one's work and having difficulty leaving it, such that time passes quickly and there is forgetfulness of everything else around. The higher the score, the higher the level of work engagement.
Balance Between Risks and Resources | 3 months
  The balance between risks and resources was measured via the BR scale developed by Mikolajczak & Roskam (2018). This scale measures the balance between the risks and resources that people have in their role as a parent. Each item is responded in a bipolar scale from -5 to +5 (going through 0). The negative pole represents a risk, while the positive pole represents a resource. A global score is composed by adding 39 items, with negative scores indicating a larger presence of risks and positive scores indicating a larger presence of resources. Moreover, each of the 39 items can be categorized as either a "common" or "specific" antecedent to parental burnout. There are 14 common antecedents and refer to general variables that could enhance parental burnout, such as finding it difficult to reconcile family and professional life. In turn, there are 15 specific antecedents to parental burnout, such as feeling that one does not have the competencies to be a good parent.
Balance Between Risks and Resources | 6 months
  The balance between risks and resources was measured via the BR scale developed by Mikolajczak & Roskam (2018). This scale measures the balance between the risks and resources that people have in their role as a parent. Each item is responded in a bipolar scale from -5 to +5 (going through 0). The negative pole represents a risk, while the positive pole represents a resource. A global score is composed by adding 39 items, with negative scores indicating a larger presence of risks and positive scores indicating a larger presence of resources. Moreover, each of the 39 items can be categorized as either a "common" or "specific" antecedent to parental burnout. There are 14 common antecedents and refer to general variables that could enhance parental burnout, such as finding it difficult to reconcile family and professional life. In turn, there are 15 specific antecedents to parental burnout, such as feeling that one does not have the competencies to be a good parent.
Balance Between Risks and Resources | 9 months
  The balance between risks and resources was measured via the BR scale developed by Mikolajczak & Roskam (2018). This scale measures the balance between the risks and resources that people have in their role as a parent. Each item is responded in a bipolar scale from -5 to +5 (going through 0). The negative pole represents a risk, while the positive pole represents a resource. A global score is composed by adding 39 items, with negative scores indicating a larger presence of risks and positive scores indicating a larger presence of resources. Moreover, each of the 39 items can be categorized as either a "common" or "specific" antecedent to parental burnout. There are 14 common antecedents and refer to general variables that could enhance parental burnout, such as finding it difficult to reconcile family and professional life. In turn, there are 15 specific antecedents to parental burnout, such as feeling that one does not have the competencies to be a good parent.
General Health | 3 months
  To measure general health, we used a scale called EQ-5D (Olivares-Tirado, 2006), which is commonly used in Chile to assess the impact of health-related interventions. This scale looks at five areas of health: mobility, personal care, ability to do regular activities (e.g., work, study, etc.), physical pain, and anxiety/depression. For each area, participants chose from three options that indicate how much difficulty they have: no difficulty, some difficulty, or unable to do it. Each option was given a score from 0 to 2, with 0 meaning no problems and 2 meaning a lot of problems.
General Health | 6 months
  To measure general health, we used a scale called EQ-5D (Olivares-Tirado, 2006), which is commonly used in Chile to assess the impact of health-related interventions. This scale looks at five areas of health: mobility, personal care, ability to do regular activities (e.g., work, study, etc.), physical pain, and anxiety/depression. For each area, participants chose from three options that indicate how much difficulty they have: no difficulty, some difficulty, or unable to do it. Each option was given a score from 0 to 2, with 0 meaning no problems and 2 meaning a lot of problems.
General Health | 9 months
  To measure general health, we used a scale called EQ-5D (Olivares-Tirado, 2006), which is commonly used in Chile to assess the impact of health-related interventions. This scale looks at five areas of health: mobility, personal care, ability to do regular activities (e.g., work, study, etc.), physical pain, and anxiety/depression. For each area, participants chose from three options that indicate how much difficulty they have: no difficulty, some difficulty, or unable to do it. Each option was given a score from 0 to 2, with 0 meaning no problems and 2 meaning a lot of problems.
General Health | 12 months
  To measure general health, we used a scale called EQ-5D (Olivares-Tirado, 2006), which is commonly used in Chile to assess the impact of health-related interventions. This scale looks at five areas of health: mobility, personal care, ability to do regular activities (e.g., work, study, etc.), physical pain, and anxiety/depression. For each area, participants chose from three options that indicate how much difficulty they have: no difficulty, some difficulty, or unable to do it. Each option was given a score from 0 to 2, with 0 meaning no problems and 2 meaning a lot of problems.
General Health | 18 months
  To measure general health, we used a scale called EQ-5D (Olivares-Tirado, 2006), which is commonly used in Chile to assess the impact of health-related interventions. This scale looks at five areas of health: mobility, personal care, ability to do regular activities (e.g., work, study, etc.), physical pain, and anxiety/depression. For each area, participants chose from three options that indicate how much difficulty they have: no difficulty, some difficulty, or unable to do it. Each option was given a score from 0 to 2, with 0 meaning no problems and 2 meaning a lot of problems.
General Health | 24 months
  To measure general health, we used a scale called EQ-5D (Olivares-Tirado, 2006), which is commonly used in Chile to assess the impact of health-related interventions. This scale looks at five areas of health: mobility, personal care, ability to do regular activities (e.g., work, study, etc.), physical pain, and anxiety/depression. For each area, participants chose from three options that indicate how much difficulty they have: no difficulty, some difficulty, or unable to do it. Each option was given a score from 0 to 2, with 0 meaning no problems and 2 meaning a lot of problems.
Burnout | 3 months
  For burnout we only used the emotional exhaustion scale translated by Olivares-Faúndez and colleagues (2014). Emotional exhaustion is composed of 7 items responded with a 5-point Likert scale representing the extent to which participants agree or disagree with a series of statement about their work. This scale measures the extent to which people feel emotionally exhausted and drained by their work, and high scores represent high levels of burnout. Example items are the extent to which participants feel "emotional drained at work", "that they are working too much", and "completely worn out at the end of the day".
Burnout | 6 months
  For burnout we only used the emotional exhaustion scale translated by Olivares-Faúndez and colleagues (2014). Emotional exhaustion is composed of 7 items responded with a 5-point Likert scale representing the extent to which participants agree or disagree with a series of statement about their work. This scale measures the extent to which people feel emotionally exhausted and drained by their work, and high scores represent high levels of burnout. Example items are the extent to which participants feel "emotional drained at work", "that they are working too much", and "completely worn out at the end of the day".
Burnout | 9 months
  For burnout we only used the emotional exhaustion scale translated by Olivares-Faúndez and colleagues (2014). Emotional exhaustion is composed of 7 items responded with a 5-point Likert scale representing the extent to which participants agree or disagree with a series of statement about their work. This scale measures the extent to which people feel emotionally exhausted and drained by their work, and high scores represent high levels of burnout. Example items are the extent to which participants feel "emotional drained at work", "that they are working too much", and "completely worn out at the end of the day".
Burnout | 12 months
  For burnout we only used the emotional exhaustion scale translated by Olivares-Faúndez and colleagues (2014). Emotional exhaustion is composed of 7 items responded with a 5-point Likert scale representing the extent to which participants agree or disagree with a series of statement about their work. This scale measures the extent to which people feel emotionally exhausted and drained by their work, and high scores represent high levels of burnout. Example items are the extent to which participants feel "emotional drained at work", "that they are working too much", and "completely worn out at the end of the day".
Burnout | 18 months
  For burnout we only used the emotional exhaustion scale translated by Olivares-Faúndez and colleagues (2014). Emotional exhaustion is composed of 7 items responded with a 5-point Likert scale representing the extent to which participants agree or disagree with a series of statement about their work. This scale measures the extent to which people feel emotionally exhausted and drained by their work, and high scores represent high levels of burnout. Example items are the extent to which participants feel "emotional drained at work", "that they are working too much", and "completely worn out at the end of the day".
Burnout | 24 months
  For burnout we only used the emotional exhaustion scale translated by Olivares-Faúndez and colleagues (2014). Emotional exhaustion is composed of 7 items responded with a 5-point Likert scale representing the extent to which participants agree or disagree with a series of statement about their work. This scale measures the extent to which people feel emotionally exhausted and drained by their work, and high scores represent high levels of burnout. Example items are the extent to which participants feel "emotional drained at work", "that they are working too much", and "completely worn out at the end of the day".
Decentering | 3 months
  scale. The scale has 11 items, responded with a 5-point Likert scale representing the extent to which participants agree or disagree with a series of statements about themselves. Higher values denote higher levels of decentering. This scale measures the extent to which participants can detach themselves from their own thoughts and experiences, and observe them from afar. Example items are: "I am able to accept myself", "I can slow my thoughts down in moments of stress", and "I can observe unpleasant feelings without being dragged into them".
Decentering | 6 months
  scale. The scale has 11 items, responded with a 5-point Likert scale representing the extent to which participants agree or disagree with a series of statements about themselves. Higher values denote higher levels of decentering. This scale measures the extent to which participants can detach themselves from their own thoughts and experiences, and observe them from afar. Example items are: "I am able to accept myself", "I can slow my thoughts down in moments of stress", and "I can observe unpleasant feelings without being dragged into them".
Decentering | 9 months
  scale. The scale has 11 items, responded with a 5-point Likert scale representing the extent to which participants agree or disagree with a series of statements about themselves. Higher values denote higher levels of decentering. This scale measures the extent to which participants can detach themselves from their own thoughts and experiences, and observe them from afar. Example items are: "I am able to accept myself", "I can slow my thoughts down in moments of stress", and "I can observe unpleasant feelings without being dragged into them".
Decentering | 12 months
  scale. The scale has 11 items, responded with a 5-point Likert scale representing the extent to which participants agree or disagree with a series of statements about themselves. Higher values denote higher levels of decentering. This scale measures the extent to which participants can detach themselves from their own thoughts and experiences, and observe them from afar. Example items are: "I am able to accept myself", "I can slow my thoughts down in moments of stress", and "I can observe unpleasant feelings without being dragged into them".
Decentering | 18 months
  scale. The scale has 11 items, responded with a 5-point Likert scale representing the extent to which participants agree or disagree with a series of statements about themselves. Higher values denote higher levels of decentering. This scale measures the extent to which participants can detach themselves from their own thoughts and experiences, and observe them from afar. Example items are: "I am able to accept myself", "I can slow my thoughts down in moments of stress", and "I can observe unpleasant feelings without being dragged into them".
Decentering | 24 months
  scale. The scale has 11 items, responded with a 5-point Likert scale representing the extent to which participants agree or disagree with a series of statements about themselves. Higher values denote higher levels of decentering. This scale measures the extent to which participants can detach themselves from their own thoughts and experiences, and observe them from afar. Example items are: "I am able to accept myself", "I can slow my thoughts down in moments of stress", and "I can observe unpleasant feelings without being dragged into them".
Emotional Regulation | 3 months
  We used a Spanish version of a scale to measure emotional regulation Cabello et al., 2013), which has two dimensions: cognitive change and suppression. Cognitive change is measured with 6 items that ask how much participants change their thinking to improve their mood. Suppression is measured with 4 items that ask how much participants control their emotions by not expressing them. Both dimensions use a 5-point Likert scale to rate agreement with statements about themselves. Higher scores indicate more cognitive change or suppression. Example items include "I control my emotions by changing my way of thinking about the situation I am in" for cognitive change and "I keep my emotions to myself" for suppression.
Emotional Regulation | 6 months
  We used a Spanish version of a scale to measure emotional regulation Cabello et al., 2013), which has two dimensions: cognitive change and suppression. Cognitive change is measured with 6 items that ask how much participants change their thinking to improve their mood. Suppression is measured with 4 items that ask how much participants control their emotions by not expressing them. Both dimensions use a 5-point Likert scale to rate agreement with statements about themselves. Higher scores indicate more cognitive change or suppression. Example items include "I control my emotions by changing my way of thinking about the situation I am in" for cognitive change and "I keep my emotions to myself" for suppression.
Emotional Regulation | 9 months
  We used a Spanish version of a scale to measure emotional regulation Cabello et al., 2013), which has two dimensions: cognitive change and suppression. Cognitive change is measured with 6 items that ask how much participants change their thinking to improve their mood. Suppression is measured with 4 items that ask how much participants control their emotions by not expressing them. Both dimensions use a 5-point Likert scale to rate agreement with statements about themselves. Higher scores indicate more cognitive change or suppression. Example items include "I control my emotions by changing my way of thinking about the situation I am in" for cognitive change and "I keep my emotions to myself" for suppression.
Emotional Regulation | 12 months
  We used a Spanish version of a scale to measure emotional regulation Cabello et al., 2013), which has two dimensions: cognitive change and suppression. Cognitive change is measured with 6 items that ask how much participants change their thinking to improve their mood. Suppression is measured with 4 items that ask how much participants control their emotions by not expressing them. Both dimensions use a 5-point Likert scale to rate agreement with statements about themselves. Higher scores indicate more cognitive change or suppression. Example items include "I control my emotions by changing my way of thinking about the situation I am in" for cognitive change and "I keep my emotions to myself" for suppression.
Emotional Regulation | 18 months
  We used a Spanish version of a scale to measure emotional regulation Cabello et al., 2013), which has two dimensions: cognitive change and suppression. Cognitive change is measured with 6 items that ask how much participants change their thinking to improve their mood. Suppression is measured with 4 items that ask how much participants control their emotions by not expressing them. Both dimensions use a 5-point Likert scale to rate agreement with statements about themselves. Higher scores indicate more cognitive change or suppression. Example items include "I control my emotions by changing my way of thinking about the situation I am in" for cognitive change and "I keep my emotions to myself" for suppression.
Emotional Regulation | 24 months
  We used a Spanish version of a scale to measure emotional regulation Cabello et al., 2013), which has two dimensions: cognitive change and suppression. Cognitive change is measured with 6 items that ask how much participants change their thinking to improve their mood. Suppression is measured with 4 items that ask how much participants control their emotions by not expressing them. Both dimensions use a 5-point Likert scale to rate agreement with statements about themselves. Higher scores indicate more cognitive change or suppression. Example items include "I control my emotions by changing my way of thinking about the situation I am in" for cognitive change and "I keep my emotions to myself" for suppression.
Personality | 3 months
  We used a Spanish version of a Big-Five scale to measure personality (Ortet et al., 2020). Although the Big-Five comprises 5 dimensions, we used only two: extraversion and neuroticism. Extraversion is measured with 6 items that ask participants the extent to which they are extraverted, assertive, and sociable. Neuroticism is measured with 6 items that ask participants the extent to which they tend to worry too much and tend to get depressed easily. Both dimensions use a 5-point Likert scale to rate agreement with statements about themselves. Higher scores indicate more extraversion and neuroticism. Example items are "I am extraverted, sociable" for extraversion and "I worry too much" for neuroticism.
Personality | 6 months
  We used a Spanish version of a Big-Five scale to measure personality (Ortet et al., 2020). Although the Big-Five comprises 5 dimensions, we used only two: extraversion and neuroticism. Extraversion is measured with 6 items that ask participants the extent to which they are extraverted, assertive, and sociable. Neuroticism is measured with 6 items that ask participants the extent to which they tend to worry too much and tend to get depressed easily. Both dimensions use a 5-point Likert scale to rate agreement with statements about themselves. Higher scores indicate more extraversion and neuroticism. Example items are "I am extraverted, sociable" for extraversion and "I worry too much" for neuroticism.
Personality | 9 months
  We used a Spanish version of a Big-Five scale to measure personality (Ortet et al., 2020). Although the Big-Five comprises 5 dimensions, we used only two: extraversion and neuroticism. Extraversion is measured with 6 items that ask participants the extent to which they are extraverted, assertive, and sociable. Neuroticism is measured with 6 items that ask participants the extent to which they tend to worry too much and tend to get depressed easily. Both dimensions use a 5-point Likert scale to rate agreement with statements about themselves. Higher scores indicate more extraversion and neuroticism. Example items are "I am extraverted, sociable" for extraversion and "I worry too much" for neuroticism.
Personality | 12 months
  We used a Spanish version of a Big-Five scale to measure personality (Ortet et al., 2020). Although the Big-Five comprises 5 dimensions, we used only two: extraversion and neuroticism. Extraversion is measured with 6 items that ask participants the extent to which they are extraverted, assertive, and sociable. Neuroticism is measured with 6 items that ask participants the extent to which they tend to worry too much and tend to get depressed easily. Both dimensions use a 5-point Likert scale to rate agreement with statements about themselves. Higher scores indicate more extraversion and neuroticism. Example items are "I am extraverted, sociable" for extraversion and "I worry too much" for neuroticism.
Personality | 18 months
  We used a Spanish version of a Big-Five scale to measure personality (Ortet et al., 2020). Although the Big-Five comprises 5 dimensions, we used only two: extraversion and neuroticism. Extraversion is measured with 6 items that ask participants the extent to which they are extraverted, assertive, and sociable. Neuroticism is measured with 6 items that ask participants the extent to which they tend to worry too much and tend to get depressed easily. Both dimensions use a 5-point Likert scale to rate agreement with statements about themselves. Higher scores indicate more extraversion and neuroticism. Example items are "I am extraverted, sociable" for extraversion and "I worry too much" for neuroticism.
Personality | 24 months
  We used a Spanish version of a Big-Five scale to measure personality (Ortet et al., 2020). Although the Big-Five comprises 5 dimensions, we used only two: extraversion and neuroticism. Extraversion is measured with 6 items that ask participants the extent to which they are extraverted, assertive, and sociable. Neuroticism is measured with 6 items that ask participants the extent to which they tend to worry too much and tend to get depressed easily. Both dimensions use a 5-point Likert scale to rate agreement with statements about themselves. Higher scores indicate more extraversion and neuroticism. Example items are "I am extraverted, sociable" for extraversion and "I worry too much" for neuroticism.
Job Resources | 3 months
  Job resources represent characteristic of the job that allow employees to cope with demands and help them flourish in their jobs. To evaluate job resources, we employed the Psychosocial Factors Questionnaire (PSF-Q75), which was validated in Spanish by Madrid and colleagues (2020). From the range of available resources, we selected three to assess, specifically, task autonomy (three items), social support (six items), and significance (three items). Our aim in choosing these resources was to represent three distinct categories of job resources, namely, task resources (autonomy), social resources (social support), and job meaning (significance). The questionnaire employed a 5-point Likert scale, which asked participants to indicate the extent to which they agreed or disagreed with various statements about their jobs. Higher scores indicated greater levels of job resources.
Job Resources | 6 months
  Job resources represent characteristic of the job that allow employees to cope with demands and help them flourish in their jobs. To evaluate job resources, we employed the Psychosocial Factors Questionnaire (PSF-Q75), which was validated in Spanish by Madrid and colleagues (2020). From the range of available resources, we selected three to assess, specifically, task autonomy (three items), social support (six items), and significance (three items). Our aim in choosing these resources was to represent three distinct categories of job resources, namely, task resources (autonomy), social resources (social support), and job meaning (significance). The questionnaire employed a 5-point Likert scale, which asked participants to indicate the extent to which they agreed or disagreed with various statements about their jobs. Higher scores indicated greater levels of job resources.
Job Resources | 9 months
  Job resources represent characteristic of the job that allow employees to cope with demands and help them flourish in their jobs. To evaluate job resources, we employed the Psychosocial Factors Questionnaire (PSF-Q75), which was validated in Spanish by Madrid and colleagues (2020). From the range of available resources, we selected three to assess, specifically, task autonomy (three items), social support (six items), and significance (three items). Our aim in choosing these resources was to represent three distinct categories of job resources, namely, task resources (autonomy), social resources (social support), and job meaning (significance). The questionnaire employed a 5-point Likert scale, which asked participants to indicate the extent to which they agreed or disagreed with various statements about their jobs. Higher scores indicated greater levels of job resources.
Job Resources | 12 months
  Job resources represent characteristic of the job that allow employees to cope with demands and help them flourish in their jobs. To evaluate job resources, we employed the Psychosocial Factors Questionnaire (PSF-Q75), which was validated in Spanish by Madrid and colleagues (2020). From the range of available resources, we selected three to assess, specifically, task autonomy (three items), social support (six items), and significance (three items). Our aim in choosing these resources was to represent three distinct categories of job resources, namely, task resources (autonomy), social resources (social support), and job meaning (significance). The questionnaire employed a 5-point Likert scale, which asked participants to indicate the extent to which they agreed or disagreed with various statements about their jobs. Higher scores indicated greater levels of job resources.
Job Resources | 18 months
  Job resources represent characteristic of the job that allow employees to cope with demands and help them flourish in their jobs. To evaluate job resources, we employed the Psychosocial Factors Questionnaire (PSF-Q75), which was validated in Spanish by Madrid and colleagues (2020). From the range of available resources, we selected three to assess, specifically, task autonomy (three items), social support (six items), and significance (three items). Our aim in choosing these resources was to represent three distinct categories of job resources, namely, task resources (autonomy), social resources (social support), and job meaning (significance). The questionnaire employed a 5-point Likert scale, which asked participants to indicate the extent to which they agreed or disagreed with various statements about their jobs. Higher scores indicated greater levels of job resources.
Job Resources | 24 months
  Job resources represent characteristic of the job that allow employees to cope with demands and help them flourish in their jobs. To evaluate job resources, we employed the Psychosocial Factors Questionnaire (PSF-Q75), which was validated in Spanish by Madrid and colleagues (2020). From the range of available resources, we selected three to assess, specifically, task autonomy (three items), social support (six items), and significance (three items). Our aim in choosing these resources was to represent three distinct categories of job resources, namely, task resources (autonomy), social resources (social support), and job meaning (significance). The questionnaire employed a 5-point Likert scale, which asked participants to indicate the extent to which they agreed or disagreed with various statements about their jobs. Higher scores indicated greater levels of job resources.
Challenge Demands | 3 months
  Challenge demands are job-related obstacles that require effort to overcome and achieve good performance. Crucially, these demands are an inherent and essential aspect of the job. To evaluate challenge demands, we employed the Spanish version of the Job Characteristics Questionnaire, which was validated by Bayona and colleagues (2015). We specifically focused on three distinct challenge demands, namely workload (six items), job complexity (four items), and information processing requirements (five items). The questionnaire utilized a 5-point Likert scale, which asked participants to indicate the extent to which they agreed or disagreed with various statements about their jobs. Higher scores indicated greater levels of challenge demands. Sample items included "I have to work very quickly" for workload, "My job requires me to work on problems that have no clear solution" for job complexity, and "My job necessitates managing a large volume of information" for information processing.
Challenge Demands | 6 months
  Challenge demands are job-related obstacles that require effort to overcome and achieve good performance. Crucially, these demands are an inherent and essential aspect of the job. To evaluate challenge demands, we employed the Spanish version of the Job Characteristics Questionnaire, which was validated by Bayona and colleagues (2015). We specifically focused on three distinct challenge demands, namely workload (six items), job complexity (four items), and information processing requirements (five items). The questionnaire utilized a 5-point Likert scale, which asked participants to indicate the extent to which they agreed or disagreed with various statements about their jobs. Higher scores indicated greater levels of challenge demands. Sample items included "I have to work very quickly" for workload, "My job requires me to work on problems that have no clear solution" for job complexity, and "My job necessitates managing a large volume of information" for information processing.
Challenge Demands | 9 months
  Challenge demands are job-related obstacles that require effort to overcome and achieve good performance. Crucially, these demands are an inherent and essential aspect of the job. To evaluate challenge demands, we employed the Spanish version of the Job Characteristics Questionnaire, which was validated by Bayona and colleagues (2015). We specifically focused on three distinct challenge demands, namely workload (six items), job complexity (four items), and information processing requirements (five items). The questionnaire utilized a 5-point Likert scale, which asked participants to indicate the extent to which they agreed or disagreed with various statements about their jobs. Higher scores indicated greater levels of challenge demands. Sample items included "I have to work very quickly" for workload, "My job requires me to work on problems that have no clear solution" for job complexity, and "My job necessitates managing a large volume of information" for information processing.
Challenge Demands | 12 months
  Challenge demands are job-related obstacles that require effort to overcome and achieve good performance. Crucially, these demands are an inherent and essential aspect of the job. To evaluate challenge demands, we employed the Spanish version of the Job Characteristics Questionnaire, which was validated by Bayona and colleagues (2015). We specifically focused on three distinct challenge demands, namely workload (six items), job complexity (four items), and information processing requirements (five items). The questionnaire utilized a 5-point Likert scale, which asked participants to indicate the extent to which they agreed or disagreed with various statements about their jobs. Higher scores indicated greater levels of challenge demands. Sample items included "I have to work very quickly" for workload, "My job requires me to work on problems that have no clear solution" for job complexity, and "My job necessitates managing a large volume of information" for information processing.
Challenge Demands | 18 months
  Challenge demands are job-related obstacles that require effort to overcome and achieve good performance. Crucially, these demands are an inherent and essential aspect of the job. To evaluate challenge demands, we employed the Spanish version of the Job Characteristics Questionnaire, which was validated by Bayona and colleagues (2015). We specifically focused on three distinct challenge demands, namely workload (six items), job complexity (four items), and information processing requirements (five items). The questionnaire utilized a 5-point Likert scale, which asked participants to indicate the extent to which they agreed or disagreed with various statements about their jobs. Higher scores indicated greater levels of challenge demands. Sample items included "I have to work very quickly" for workload, "My job requires me to work on problems that have no clear solution" for job complexity, and "My job necessitates managing a large volume of information" for information processing.
Challenge Demands | 24 months
  Challenge demands are job-related obstacles that require effort to overcome and achieve good performance. Crucially, these demands are an inherent and essential aspect of the job. To evaluate challenge demands, we employed the Spanish version of the Job Characteristics Questionnaire, which was validated by Bayona and colleagues (2015). We specifically focused on three distinct challenge demands, namely workload (six items), job complexity (four items), and information processing requirements (five items). The questionnaire utilized a 5-point Likert scale, which asked participants to indicate the extent to which they agreed or disagreed with various statements about their jobs. Higher scores indicated greater levels of challenge demands. Sample items included "I have to work very quickly" for workload, "My job requires me to work on problems that have no clear solution" for job complexity, and "My job necessitates managing a large volume of information" for information processing.
Hindrance Demands | 3 months
  Hindrance demands refer to job-related obstacles that hinder work performance. Unlike challenge demands, hindrance demands are usually not inherent to the job itself. To measure hindrance demands, we utilized the Questionnaire on the Experience and Assessment of Work, developed by Van Veldhoven and Meijman (1994). We selected three typical hindrance demands that workers encounter, namely interdependence (three items), emotional demands (five items), and role conflict (four items). The questionnaire employed a 5-point Likert scale that required participants to indicate the extent to which they agreed or disagreed with various statements related to their jobs. Higher scores represented greater levels of hindrance demands. Sample items included "I cannot finish my job until others complete theirs" for interdependence, "My job is often emotionally draining" for emotional demands, and "I am required to perform contradictory tasks at work" for role conflict.
Hindrance Demands | 6 months
  Hindrance demands refer to job-related obstacles that hinder work performance. Unlike challenge demands, hindrance demands are usually not inherent to the job itself. To measure hindrance demands, we utilized the Questionnaire on the Experience and Assessment of Work, developed by Van Veldhoven and Meijman (1994). We selected three typical hindrance demands that workers encounter, namely interdependence (three items), emotional demands (five items), and role conflict (four items). The questionnaire employed a 5-point Likert scale that required participants to indicate the extent to which they agreed or disagreed with various statements related to their jobs. Higher scores represented greater levels of hindrance demands. Sample items included "I cannot finish my job until others complete theirs" for interdependence, "My job is often emotionally draining" for emotional demands, and "I am required to perform contradictory tasks at work" for role conflict.
Hindrance Demands | 9 months
  Hindrance demands refer to job-related obstacles that hinder work performance. Unlike challenge demands, hindrance demands are usually not inherent to the job itself. To measure hindrance demands, we utilized the Questionnaire on the Experience and Assessment of Work, developed by Van Veldhoven and Meijman (1994). We selected three typical hindrance demands that workers encounter, namely interdependence (three items), emotional demands (five items), and role conflict (four items). The questionnaire employed a 5-point Likert scale that required participants to indicate the extent to which they agreed or disagreed with various statements related to their jobs. Higher scores represented greater levels of hindrance demands. Sample items included "I cannot finish my job until others complete theirs" for interdependence, "My job is often emotionally draining" for emotional demands, and "I am required to perform contradictory tasks at work" for role conflict.
Hindrance Demands | 12 months
  Hindrance demands refer to job-related obstacles that hinder work performance. Unlike challenge demands, hindrance demands are usually not inherent to the job itself. To measure hindrance demands, we utilized the Questionnaire on the Experience and Assessment of Work, developed by Van Veldhoven and Meijman (1994). We selected three typical hindrance demands that workers encounter, namely interdependence (three items), emotional demands (five items), and role conflict (four items). The questionnaire employed a 5-point Likert scale that required participants to indicate the extent to which they agreed or disagreed with various statements related to their jobs. Higher scores represented greater levels of hindrance demands. Sample items included "I cannot finish my job until others complete theirs" for interdependence, "My job is often emotionally draining" for emotional demands, and "I am required to perform contradictory tasks at work" for role conflict.
Hindrance Demands | 18 months
  Hindrance demands refer to job-related obstacles that hinder work performance. Unlike challenge demands, hindrance demands are usually not inherent to the job itself. To measure hindrance demands, we utilized the Questionnaire on the Experience and Assessment of Work, developed by Van Veldhoven and Meijman (1994). We selected three typical hindrance demands that workers encounter, namely interdependence (three items), emotional demands (five items), and role conflict (four items). The questionnaire employed a 5-point Likert scale that required participants to indicate the extent to which they agreed or disagreed with various statements related to their jobs. Higher scores represented greater levels of hindrance demands. Sample items included "I cannot finish my job until others complete theirs" for interdependence, "My job is often emotionally draining" for emotional demands, and "I am required to perform contradictory tasks at work" for role conflict.
Hindrance Demands | 24 months
  Hindrance demands refer to job-related obstacles that hinder work performance. Unlike challenge demands, hindrance demands are usually not inherent to the job itself. To measure hindrance demands, we utilized the Questionnaire on the Experience and Assessment of Work, developed by Van Veldhoven and Meijman (1994). We selected three typical hindrance demands that workers encounter, namely interdependence (three items), emotional demands (five items), and role conflict (four items). The questionnaire employed a 5-point Likert scale that required participants to indicate the extent to which they agreed or disagreed with various statements related to their jobs. Higher scores represented greater levels of hindrance demands. Sample items included "I cannot finish my job until others complete theirs" for interdependence, "My job is often emotionally draining" for emotional demands, and "I am required to perform contradictory tasks at work" for role conflict.
Microbiota | 3 months
  Genomic DNA from fecal samples, with a focus on 16s ribosomal RNA. It will be measured only in a subgroup of 32 participants from both the intervention arm (n=16) and the active control arm (n=16).
Microbiota | 6 months
  Genomic DNA from fecal samples, with a focus on 16s ribosomal RNA. It will be measured only in a subgroup of 32 participants from both the intervention arm (n=16) and the active control arm (n=16).
Respiratory sinus arrhythmias | 3 months
  Simultaneously, the synchronization between heart rate variability and respiratory rate will be studied, filtering both signals to eliminate artifacts. Respiratory sinus arrhythmias will be analyzed as an indirect indicator of vagal tone. It will be measured only in a subgroup of 32 participants from both the intervention arm (n=16) and the active control arm (n=16).
Respiratory sinus arrhythmias | 6 months
  Simultaneously, the synchronization between heart rate variability and respiratory rate will be studied, filtering both signals to eliminate artifacts. Respiratory sinus arrhythmias will be analyzed as an indirect indicator of vagal tone. It will be measured only in a subgroup of 32 participants from both the intervention arm (n=16) and the active control arm (n=16).

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier VILLALON LOPEZ, Principal Investigator — Diego Portales University
Locations (1):
- University Diego Portales, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided